CLINICAL TRIAL: NCT04089085
Title: STRONGer Together: A Small Group Intervention for Children With Asthma and Anxiety/Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: Sigma Theta Tau International (Other)
Responsible Party: Principal Investigator, Colleen McGovern, Assistant Professor, University of North Carolina, Greensboro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-1290
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Childhood Asthma; Childhood Anxiety; Childhood Depression
Keywords: Childhood Asthma; Childhood Anxiety/depression; Educational and Behavioral Intervention for Children
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: One Group Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group pilot (Other): The experimental group will receive the intervention, which is an 8-week (30 minute session per week) asthma educational and cognitive behavioral skills program.
  Interventions: Behavioral: STRONGer Together

INTERVENTIONS:
Behavioral: STRONGer Together — STRONGer (Successes/Strengths, Triggers, Remember your medications, Ongoing communication, Never give up!, Gratitude) Together is an asthma educational and cognitive behavioral skills intervention for children between 8 - 12 years of age. The intervention is implemented in small groups in 30-minute sessions.

SUMMARY:
The proposed study is a one group pilot to assess the feasibility and acceptability of an 8-session intervention (STRONGer Together) for children between 8 - 12 years of age with asthma and anxiety/depressive symptoms.

DETAILED DESCRIPTION:
Asthma is one of the leading chronic conditions in children and affects 6.1 million children in the United States. 5,15,16 It is one of the most common causes of school absenteeism and is a major public health issue, accounting for over $56 billion dollars annually in healthcare costs. 16 Children with asthma have increased odds ~ 3.13 of having co-morbid anxiety/depression, a lower quality of life, and higher morbidity and mortality rates. 4,17-21 In recent years, the economic burden of asthma 22 and the level of impairment due to mental health concerns have increased for children and adolescents. 23 A study by Secinti, Thompson, Richards, and Gaysina (2017) highlights the association between childhood chronic physical conditions and adult emotional health, further emphasizing the critical need to address physical health as well as the emotional and mental health of children with asthma. 24 More distally, asthma, anxiety, and depression cause inflammation. 25 Left unaddressed, adults with asthma and comorbid anxiety/depression may be at higher risk of cardiovascular disease. 25,26 Compounding potential health related complications of asthma and comorbid anxiety/depressive symptoms is the disproportionate effect of asthma for children from ethnic and racial minority populations 4,19 or from socioeconomically disadvantaged settings. 19 Further, underserved populations are less likely to receive appropriate medical or mental health care for a variety of reasons such as transportation, neighborhood factors, a caregiver's inability to pay for needed medications or treatment, and healthcare provider bias. 20 Cost-related barriers were found to be most indicative of uncontrolled asthma in a recent study. 27 Clinicians, policy makers, and researchers must be responsive and provide interventions to ameliorate detrimental outcomes. Prior studies indicate that not only are children with asthma and anxiety/depression less likely to adhere to treatment guidelines, they are prone to misinterpretation of their symptoms leading to overuse of their quick-relief inhaler. 20 Symptoms of anxiety and asthma are often confused and psychological factors can be a trigger for an asthma attack. 25 Improvement in symptom interpretation, asthma self-efficacy, and asthma illness beliefs has been associated with better asthma control. 28 Children using skills to take care of their asthma, or asthma self-management, is a dynamic process. Self-efficacy contributes to one's to self-management behaviors. 29 While many factors contribute to managing one's asthma, the skills can be easily learned. However, children with asthma are frequently expected to manage their medications at a very young age and may not have the knowledge or skills yet to understand what actions to take and when. For example, a study by Orrell-Valente, Jarlsberg, Hill, and Cabana (2008) found that 20% of children aged 7 years were responsible for managing their asthma medications, and by age 11 years, 50% of children are left to manage their asthma medications without caregiver assistance. 30 Bellin and colleagues (2017) interviewed children as young as six years of age that self-administered their medication. 31 Because of this, educating children about asthma is imperative so they can more accurately interpret their symptoms and treat themselves for optimal health, particularly since it is a lifelong condition. The proposed one group pilot will determine the feasibility and acceptability of an 8-session educational and skills-building intervention in YMCA after-school programs in Orange and Chatham counties, and one school in Durham county in North Carolina.

ELIGIBILITY:
Inclusion Criteria:

* In the range of 8 - 12 years of age,
* Child has a diagnosis of asthma or reactive airway and prescribed a controller medication or have intermittent symptoms,
* Child has at least slightly elevated anxiety or depressive symptoms upon screening at enrollment,
* The parent/caregiver can understand and answer the survey questions in English; child can understand English in a small group setting and can answer survey questions in English,
* The consenting parent/caregiver has at least equal responsibility for the day-to-day management of the child's asthma.

Exclusion Criteria:

* Child has other pulmonary conditions (e.g., cystic fibrosis/pulmonary fibrosis),
* Child or parent/caregiver cannot answer the survey questions due to a cognitive delay.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 8-weeks
  Feasibility will be established if 80% of the participants attend 6 out of 8 sessions.
Acceptability related to the Intervention | 8 weeks
  Acceptability will be established if 80% of the child participants practice the skills or practice sheets.
Acceptability of the Intervention - for the Child Participants | 8 weeks
  Questions relate to satisfaction with the program and general like/dislike (rated 0 - 5; higher score reflects more satisfaction) and qualitative questions about what participants liked or would change about the program.
Acceptability of the Intervention - for the Parent/Caregiver Participants | 8 weeks
  Questions relate to overall satisfaction with the program (0 - 5; higher score reflects greater satisfaction) and qualitative questions about if/what their child learned from the program.

SECONDARY OUTCOMES:
Asthma Management Self-Efficacy - Child | From baseline to post-intervention (8-weeks) and at 16 weeks post-intervention.
  The Child Asthma Self-Efficacy (CASE) scale (14 items) measures children's perception of their own ability to manage asthma (e.g., "...can tell when a serious breathing problem can be controlled at home") and assesses asthma symptoms, health status, and impact of the child's illness on the family (Bursch, Schwankovsky, Gilbert, & Zeiger, 1999). Answers are scored 1 - 5; higher scores indicate greater self-efficacy.
Anxiety Measure (Screen for Child Anxiety Related Disorders [SCARED]) - Child | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The SCARED measure assesses five factors including panic/somatic, general anxiety disorder, separation anxiety, social phobia, and school phobia; it has been validated with children and adolescents ages 8 - 19 years (Beidas et al., 2015; Hale, Crocetti, Raaijmakers, & Meeus, 2011; Birmaher et al., 1999). Items are scored from 0 (not true or hardly ever true) to 2 (very true or often true; Birmaher et al., 1999). Higher scores indicate greater anxiety with a total score of 25 as having a potential anxiety disorder and 30 as more specific.
Depression Measure (Patient-Reported Outcomes Measurement Information System [PROMIS]- Child Depression Short Form) | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The PROMIS Child Depression Short Form Assesses negative mood (e.g., sadness), decrease in positive affect (e.g., loss of interest), negative views of self (e.g., worthlessness), and negative social cognition (e.g., loneliness, interpersonal alienation; Assessment Center, n.d.). Items are scored from 0 (never) to 4 (almost always). Higher scores indicate greater depressive symptoms.
Asthma Illness Representations - Child Version (AIRS-C) | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The AIRS-C is a 17-item measure designed to identify barriers to and risk factors for under-utilization of controller medications. Higher scores indicate closer alignment with the professional model of asthma management.
Pediatric Asthma Quality of Life Questionnaire (PAQLQ) - Child | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The PAQLQ 14-item Likert-type scale is validated for children between ages 7 - 17 years (Juniper, Guyatt, Ferrie, & Griffith, 1993) and measures the functional problems (symptoms, activity limitations, emotional function) that are troublesome to children with asthma (Juniper et al., 1993). Items are scored from 1 (extremely bothered) to 7 (not bothered at all) and the total score is the mean of items. Higher scores denote better QoL.
Peak Flow - Child | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The child participants will be asked to complete peak flow assessments (blowing into the meter) during the study to evaluate lung function. A higher number indicates better lung function.
Pediatric Symptom Checklist - completed by the Parent/Caregiver | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The PSC includes 17 Likert type questions to assess internalizing, attention, and externalizing problems (Murphy et al., 2016). Items are scored from 0 (never) to 2 (often; α = .89). Examples of questions include "My child feels sad, unhappy" and "Daydreams too much." Higher scores indicate more symptoms.
Asthma Control Test - Combined Child and Parent/Caregiver | From baseline to 8 weeks (immediately post-intervention) and 16 weeks post-intervention
  The C-ACT consists of questions for children (ages 4-11 years; 4 items) and parents (3 items) and the ACT (for individuals 12 years and older) has similar questions which are self-administered. This instrument assesses interference with activities, asthma symptoms, and nighttime awakenings. The C-ACT (α = .79; Lui et al., 2007; Lui et al., 2010) classifies children as very poorly controlled, not well-controlled, or well controlled.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McGovern, PhD, Principal Investigator — University of North Carolina, Greensboro
Locations (1):
- Excelsior School, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.